CLINICAL TRIAL: NCT02690415
Title: Effect of Antibiotics on Community-Associated Staphylococcus Aureus Colonization and Recurrent Infection in Patients With Uncomplicated S. Aureus Skin Abscesses
Brief Title: Community-Assoc. S. Aureus Colonization and Recurrent Infection in Pts With Uncomplicated S. Aureus Skin Abscesses
Acronym: CIRCUS
Status: Completed | Type: Observational
Sponsor: Southern Illinois University (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: ROD-SIU-14-197-CIRCUS
Record Dates: First submitted 2016-02-11; First posted 2016-02-24 (Estimated); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: MRSA

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — colonization swabs from the nose, axilla, inguinal folds and wound isolate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Antibiotics Given: Patients who's treating physician prescribed antibiotics following incision and drainage of their abscess.
  Interventions: Procedure: Antibiotics Given; Procedure: Antibiotics not given
- Antibiotics Not Given: Patients who's treating physician did not prescribed antibiotics following incision and drainage of their abscess.
  Interventions: Procedure: Antibiotics Given; Procedure: Antibiotics not given

INTERVENTIONS:
Procedure: Antibiotics Given — Patients who's treating physician prescribed antibiotics
Procedure: Antibiotics not given — Patients who's treating physician did not prescribed antibiotics

SUMMARY:
Infections due to S. aureus are a major healthcare burden. Currently there is not an effective way to prevent S. aureus infection. Treatment failure can happen in up to 20% of patients with SSTI and mean additional cost per patient can be over $1500. Antibiotics are often prescribed for the treatment of CA-S. aureus SSTI. Current IDSA CA-MRSA guidelines suggest that incision and drainage alone may be adequate for management of uncomplicated CA-S. aureus skin abscesses and there is uncertainty about the need of antibiotics. It is not known whether antibiotics are helpful in decreasing S. aureus colonization rates or preventing future S. aureus infections. Though resolution of acute abscess after drainage may be unchanged by antibiotic administration, the impact of managing S. aureus abscess without antibiotics on ongoing S. aureus colonization and recurrent infection requires further study. This study seeks to examine whether the management of initial S. aureus abscesses with incision and drainage in addition to antibiotic therapy is an effective means of preventing recurrent infection. The prolonged longitudinal follow-up of this study is another unique characteristic that will enable the investigators to capture data about recurrences of infections.

DETAILED DESCRIPTION:
Methicillin-resistant Staphylococcus aureus (MRSA) was once associated almost exclusively with healthcare-associated infections. However, new epidemic strains have emerged outside of the healthcare environment designated community-associated (CA) MRSA. From 1999 to 2005, hospitalizations for Staphylococcus aureus-related skin and soft tissue infections (SSTI) in the United States increased 4-fold to nearly 90,000 annually. At Memorial Medical Center (MMC) Emergency Department (ED) and Express Cares (EC) there have been over 6500 visits in the last 6 years secondary to SSTI.

Current Infectious Diseases Society of America (IDSA) guidelines suggest incision and drainage alone (without antibiotics) may be adequate management for uncomplicated MRSA skin abscesses. However, patients not receiving antibiotics are more likely to develop recurrent infections, which may be a result of persistent MRSA colonization. The investigators will conduct a prospective case-control study at MMC ED, EC and MMC primary care clinics of pediatric patients with skin abscesses comparing outcomes for those who received antibiotics (cases) versus those who did not (controls). This will not be an intervention study - both surgical and medical management of patients with skin abscesses will be at the discretion of the treating physician.

The central hypothesis is that the inclusion of systemic antibiotics in the management of S. aureus skin abscesses will decrease S. aureus colonization, and subsequently the incidence of recurrent SSTI in the year following baseline infection. To gain a better understanding of this problem, the investigators propose the following specific aims:

ELIGIBILITY:
Inclusion Criteria:

* (1) Children 6 months to 18 years presenting with a skin abscess.
* (2) Positive MRSA or MSSA culture from previous or current abscess

Exclusion Criteria:

* (1) Immunodeficiency;
* (2) Hospitalization within the prior 14 days
* (3) Use of mupirocin, clorhexidine or bleach water baths in the last month
* (4) Systemic antibacterial therapy with anti-staphylococcal activity within the prior 14 days.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients presenting in the Emergency Department or Express Cares and Primary Care Clinics with skin abscesses who do and do not receive antibiotic therapy at two time points.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Determine if there is a change in colonization status from baseline | At the time of surgical incision and drainage of the baseline skin abscess and 1 month post
  To determine S. aureus colonization status at three body sites (nose, axilla and inguinal folds) in pediatric patients presenting in the Emergency Department or Express Cares and Primary Care Clinics with skin abscesses who do and do not receive antibiotic therapy at two time points.
Measure incidence of recurrent SSTI | 1, 3, 6 and 12 months
  To measure incidence of recurrent SSTI at 1, 3, 6 and 12 months in patients who did or did not receive antibiotic therapy.

SECONDARY OUTCOMES:
Measure S. aureus antibiotic resistance in patients who did and did not receive antibiotics | At the time of surgical incision and drainage of the baseline skin abscess and 1 month post

CONTACTS AND LOCATIONS:
Overall Officials: Marcela Rodriguez, MD, Principal Investigator — SIU School of Medicine
Locations (1):
- SIU School of Medicine, Springfield, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hogan, Patrick G., et al.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-09): https://cdn.clinicaltrials.gov/large-docs/15/NCT02690415/Prot_SAP_000.pdf